CLINICAL TRIAL: NCT02440711
Title: Endurance, Energy Expenditure, Perceived Function, and Satisfaction of Persons With Transtibial Limb Loss Using a Running-Specific Prosthesis Modified for Walking
Brief Title: Evaluation of a Modified Running-specific Prosthetic Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Brian Hafner, Associate Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 49150
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Transtibial Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mRSF-ESF (Experimental): Study participants in Arm 1 will first receive the Modified running specific foot (mRSF) and then the Energy storing foot (ESF). Outcomes will be assessed (in each condition) after 1 month of use. Order of interventions will be randomly assigned.
  Interventions: Device: Energy storing foot (ESF); Device: Modified running specific foot (mRSF)
- ESF-mRSF (Experimental): Study participants in Arm 2 will first receive the Energy storing foot (ESF) and then the Modified running specific foot (mRSF). Outcomes will be assessed (in each condition) after 1 month of use. Order of interventions will be randomly assigned.
  Interventions: Device: Energy storing foot (ESF); Device: Modified running specific foot (mRSF)

INTERVENTIONS:
Device: Energy storing foot (ESF) — A commercially-available energy storing prosthetic foot
  Other Names: Ossur Vari-flex
Device: Modified running specific foot (mRSF) — A running specific prosthetic foot customized for both running and walking activities
  Other Names: Ossur Cheetah (modified); Ossur Xplore

SUMMARY:
The goal of this study is to evaluate endurance, walking performance, mobility, and perceived exertion of transtibial prosthesis users (i.e., study participants) walking with a conventional energy storing prosthetic foot (ESF) and a novel modified running-specific prosthesis (mRSF). A randomized cross-over study will be conducted to determine if the mRSF provides superior performance to the ESF, which is commonly prescribed to most active individuals with lower limb amputation.

DETAILED DESCRIPTION:
Amputation of a limb is a life-altering event with profound physical, psychological, and social implications. To address their functional, vocational, and recreational needs, people with lower limb amputation (LLA) are often provided with a prosthesis or artificial leg. While use of a prosthesis can allow an individual to achieve a basic level of functional mobility, absence of an anatomical foot and ankle still impairs their physical performance. As a result, people with LLA regularly exhibit decreased walking speeds, diminished endurance, and restricted ability to participate in desired life situations.

Over the past three decades, increasingly sophisticated prosthetic foot designs have been developed by the prosthetics industry to replace amputated structures in the leg. Contemporary, energy storing feet (ESF) employ advanced materials and unique geometric designs to improve walking performance and endurance of their users. Although prosthetic limbs with ESF allow people with LLA the potential to return to an active lifestyle, even the most advanced ESF do not significantly reduce the increased energy demands required for walking when compared to conventional prosthetic feet.

Commercially-available running-specific feet (RSF) like the Össur Cheetah (Össur, Reykjavik, Iceland) allow people with LLA to participate in athletic activities and sporting events. RSF provide significantly enhanced performance, compared to traditional ESF, by extending the length and increasing the stiffness of the prosthetic keel (forefoot). RSF also do not include a heel, as they are used only for running activities. Although transtibial runners with RSF exhibit endurance levels similar to non-amputees, the RSF design does not allow the biomechanical movements or provide the stability needed to use the foot for walking (over level or uneven terrain).

A novel modified running-specific foot (mRSF) has been developed to integrate the performance of a RSF with the utility of an ESF. The mRSF combines the running keel (forefoot) of a RSF with the walking heel of a ESF. The mRSF can then be used for walking, running, and other routine daily activities. Preliminary feedback on the mRSF suggests that users experience improved overall function and high satisfaction with the device. However, empirical evidence is needed to support prescription of this prosthetic foot at other clinical facilities.

The goal of this study is therefore to evaluate endurance, walking performance, mobility, and perceived exertion of transtibial prosthesis users (i.e., study participants) walking with a conventional ESF and the mRSF. Results will be compared to determine if the mRSF provides superior performance to the ESF, which is commonly prescribed to most active individuals with LLA.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral, transtibial (below-knee) amputation from non-dysvascular causes
* Medicare functional classification level (K-level) 3 or higher (unlimited community ambulatory)
* prosthetic user for > 1 year
* scheduled to receive a mRSF prosthesis
* able and willing to participate in the study protocol (e.g., treadmill walking, overground walking, respond to survey questions, able to read and write English)

Exclusion Criteria:

* contralateral lower or upper limb involvement
* any health condition that would limit participation in the study procedures (e.g., skin breakdown, heart disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hafner, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Morgan SJ, McDonald CL, Halsne EG, Cheever SM, Salem R, Kramer PA, Hafner BJ. Laboratory- and community-based health outcomes in people with transtibial amputation using crossover and energy-storing prosthetic feet: A randomized crossover trial. PLoS One. 2018 Feb 7;13(2):e0189652. doi: 10.1371/journal.pone.0189652. eCollection 2018. PMID 29414988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 participants were screened for eligibility between May 15, 2015 and 09/26/2017 at a research laboratory in Seattle, WA.
Pre-assignment Details: 39 participants were randomized. 3 participants did not meet the eligibility criteria. 36 participants were enrolled.
Period: First Intervention
Arm/Group | mRSF-ESF | ESF-mRSF
Started | 16 | 20
Unilateral Amputation | 14 (Number of participants with unilateral amputation in the mRSF-ESF sequence to complete the first period.) | 17 (Number of participants with unilateral amputation in the ESF-mRSF sequence to complete the first period.)
Bilateral Amputation | 2 (Number of participants with bilateral amputation in the mRSF-ESF sequence to complete the first period.) | 3 (Number of participants with bilateral amputation in the ESF-mRSF sequence to complete the first period.)
Completed | 16 | 20
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | mRSF-ESF | ESF-mRSF
Started | 16 | 20
Unilateral Amputation | 14 (Number of participants with unilateral amputation in the mRSF-ESF sequence to complete the second period.) | 17 (Number of participants with unilateral amputation in the ESF-mRSF sequence to complete the second period.)
Bilateral Amputation | 2 (Number of participants with bilateral amputation in the mRSF-ESF sequence to complete the second period.) | 3 (Number of participants with bilateral amputation in the ESF-mRSF sequence to complete the second period.)
Completed | 15 | 20
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mRSF-ESF | ESF-mRSF | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 20 | 35
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (10.6) | 44.0 (11.6) | 44.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 19 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 20 | 36
Height [Mean (Standard Deviation); unit: centimeters] | 180.9 (8.6) | 176.6 (10.3) | 178.5 (9.7)
Weight [Mean (Standard Deviation); unit: kilograms] | 82.5 (12.7) | 85.9 (22.3) | 84.4 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Oxygen Consumption (VO2), Participants With Unilateral Amputation
Description: Breath-by-Breath VO2 was collected as participants walked on a treadmill at self selected fast, normal, and slow speeds. Participants walked for 6 minutes at each speed (and in each experimental condition). VO2 was normalized energy expenditure to each participant's biological mass (i.e., body mass without prosthesis) Normalized VO2 data were averaged to produce 30-s values for minutes 3-6 of each trial. These 30-s values were used in for the described analyses. Both gross and net VO2 were examined, but produced similar results, so only gross VO2 results are reported.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from 27 participants with unilateral amputation. Data from 1 participant who did not complete the protocol and 3 participants who experienced serious life events unrelated to the study that disproportionately affected one phase of the study were not analyzed.
Measure: Mean (Standard Deviation); unit: ml/min
Groups:
- mRSF (Unilateral): Participants with unilateral amputation tested while wearing the mRSF.
- ESF (Unilateral): Participants with unilateral amputation tested while wearing the ESF.
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
ml/min
  VO2 - slow walking speed | 1041.1 (246.1) | 1077.4 (245.2)
  VO2 - comfortable walking speed | 1210.9 (280.9) | 1253.5 (276.3)
  VO2 - fast walking speed | 1509.6 (398.8) | 1565.1 (376.4)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Analysis of VO2 at slow walking speed; Test type: Superiority; p = .18, Multivariate regression — A significance threshold for all analyses was set at α=0.05. Bonferroni corrections for multiple comparisons were applied; The multivariate regression included participants' biological masses and walking speeds as covariates
Statistical Analysis 2: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Analysis of VO2 at comfortable walking speed; Test type: Superiority; p = .21, Multivariate regression — [p-value comment as in outcome 1, analysis 1]; The multivariate regression included participants' biological masses and walking speeds as covariates
Statistical Analysis 3: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Analysis of VO2 at fast walking speed; Test type: Superiority; p = .16, Multivariate regression — [p-value comment as in outcome 1, analysis 1]; The multivariate regression included participants' biological masses and walking speeds as covariates

2. Primary Outcome: Metabolic Oxygen Consumption (VO2), Participants With Bilateral Amputation
Description: as for outcome 1
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: ml/min
Groups:
- mRSF (Bilateral): Participants with bilateral amputation tested while wearing the mRSF.
- ESF (Bilateral): Participants with bilateral amputation tested while wearing the ESF.
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
ml/min
  VO2 - slow walking speed | 779.6 (299.2) | 867.3 (397.7)
  VO2 - comfortable walking speed | 889.9 (300.8) | 985.0 (413.4)
  VO2 - fast walking speed | 1081.9 (319.0) | 1162.8 (439.3)

3. Primary Outcome: Six-minute Walk Test (6MWT), Participants With Unilateral Amputation
Description: Participants were asked to walk as far as possible in 6 minutes. Participants walked around cones placed 30m apart in a level hallway. Total distance (in meters) walked in 6 minutes was recorded.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
meters | 543.3 (92.6) | 537.1 (100.8)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Test type: Superiority; p = .29, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

4. Primary Outcome: Six-minute Walk Test (6MWT), Participants With Bilateral Amputation
Description: as for outcome 3
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
meters | 441.1 (72.7) | 448.9 (77.5)

5. Primary Outcome: Borg Rating of Perceived Exertion (CR100), Participants With Unilateral Amputation
Description: Participants were asked to self-report their level of perceived exertion after completing the 6MWT. Participants were shown the Borg CR100 rating scale and asked to identify their level of exertion on a scale ranging from 0 to 120. Higher scores mean greater exertion.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
units on a scale | 36.4 (31.4) | 47.3 (28.0)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Test type: Superiority; p = 0.05, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

6. Primary Outcome: Borg Rating of Perceived Exertion (CR100), Participants With Bilateral Amputation
Description: as for outcome 5
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
units on a scale | 30.4 (21.7) | 35.6 (19.2)

7. Primary Outcome: Walking Speed, Participants With Unilateral Amputation
Description: Walking speed (m/s) was assessed with a 16-foot CIR GAITRite instrumented walkway while participants performed the 6-minute walk test (6MWT).
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters / second
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
meters / second | 1.62 (0.29) | 1.60 (0.31)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Test type: Superiority; p = .25, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

8. Primary Outcome: Walking Speed, Participants With Bilateral Amputation
Description: as for outcome 7
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: meters / second
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
meters / second | 1.35 (0.23) | 1.35 (0.28)

9. Primary Outcome: Step Width, Participants With Unilateral Amputation
Description: Step width was assessed with a 16-foot CIR GAITRite instrumented walkway while participants performed the 6-minute walk test (6MWT).
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
centimeters | 13.7 (3.8) | 13.7 (3.5)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Test type: Superiority; p = .86, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

10. Primary Outcome: Step Width, Participants With Bilateral Amputation
Description: as for outcome 9
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
centimeters | 16.9 (5.4) | 16.7 (5.0)

11. Primary Outcome: Step Length, Participants With Unilateral Amputation
Description: Step length (cm) was assessed with a 16-foot CIR GAITRite instrumented walkway while participants performed the 6-minute walk test (6MWT). Step length is reported for both the prosthetic and sound (intact) limbs.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
centimeters
  Prosthetic side | 78.8 (9.2) | 79.4 (9.4)
  Sound side | 79.5 (10.2) | 76.5 (9.8)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Prosthetic side step length results; Test type: Superiority; p = .14, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05
Statistical Analysis 2: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Sound side step length results; Test type: Superiority; p < 0.001, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

12. Primary Outcome: Step Length, Participants With Bilateral Amputation
Description: as for outcome 11
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
centimeters
  Left side | 0.69 (0.08) | 0.68 (0.13)
  Right side | 0.69 (0.11) | 0.69 (0.12)

13. Primary Outcome: Step Time, Participants With Unilateral Amputation
Description: Step time was assessed with a 16-foot CIR GAITRite instrumented walkway while participants performed the 6-minute walk test (6MWT). Step time is reported for both the prosthetic and sound (intact) limbs.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
seconds
  Prosthetic side | 0.49 (0.05) | 0.49 (0.05)
  Sound side | 0.50 (0.05) | 0.50 (0.05)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Prosthetic side step time results; Test type: Superiority; p = .61, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05
Statistical Analysis 2: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Sound side step time results; Test type: Superiority; p = .40, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

14. Primary Outcome: Step Time, Participants With Bilateral Amputation
Description: as for outcome 13
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
seconds
  Right side | 0.53 (0.05) | 0.52 (0.04)
  Left side | 0.51 (0.04) | 0.51 (0.03)

15. Secondary Outcome: Daily Step Activity, Participants With Unilateral Amputation
Description: Daily step activity (steps / day) were measured over the 2-week period prior to assessment using a Orthocare Innovations Stepwatch 3 activity monitor.
Time Frame: Participants' step count data from the 2 weeks prior to in-person testing.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
steps per day | 4109 (1517) | 4307 (1750)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Test type: Superiority; p = .14, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

16. Secondary Outcome: Daily Step Activity, Participants With Bilateral Amputation
Description: as for outcome 15
Time Frame: Participants' step count data from the 2 weeks prior to in-person testing.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
steps per day | 2464 (455) | 3007 (617)

17. Secondary Outcome: Prosthetic Limb Users Survey of Mobility (PLUS-M), Participants With Unilateral Amputation
Description: The PLUS-M is a self-report instrument designed to evaluate respondent's prosthetic mobility. It is scored using a standardized T-score centered on a national sample of unilateral lower limb prosthesis users (mean = 50, standard deviation = 10). Participants were administered the PLUS-M computerized adaptive test and 12-item form on an iPad tablet. The most precise score (i.e., score with the lowest error) was used for analysis. Absolute score range from 0 to 100. Higher T-scores indicate greater mobility.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
T-score | 64.2 (7.7) | 59.3 (7.5)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Test type: Superiority; p = 0.001, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

18. Secondary Outcome: Prosthetic Limb Users Survey of Mobility (PLUS-M), Participants With Bilateral Amputation
Description: as for outcome 17
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
T-score | 59.3 (3.8) | 54.8 (6.2)

19. Secondary Outcome: Patient Reported Outcome Measurement Information System - Fatigue (PROMIS-Fatigue), Participants With Unilateral Amputation
Description: The PROMIS-Fatigue is a self-report instrument designed to evaluate respondent's symptoms and effects of fatigue. It is scored using a standardized T-score centered on the US general population (mean = 50, standard deviation = 10). Participants were administered the computerized adaptive test and a 12-item short form on an iPad tablet. The most precise score (i.e., score with the lowest error) was used for analysis. Absolute score range from 0 to 100. Higher T-scores indicate greater fatigue.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
T-score | 45.4 (7.5) | 49.1 (7.4)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Test type: Superiority; p = 0.001, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

20. Secondary Outcome: Patient Reported Outcome Measurement Information System - Fatigue (PROMIS-Fatigue), Participants With Bilateral Amputation
Description: as for outcome 19
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
T-score | 42.1 (8.9) | 47.7 (6.2)

21. Secondary Outcome: Activities-Specific Balance Confidence Scale (ABC), Participants With Unilateral Amputation
Description: The ABC is a self-report instrument designed to evaluate respondent's confidence in performing normal daily activities. It is scored from 0 to 4. Participants were administered an electronic version of the ABC on an iPad tablet. Scores range from 0 to 4. Higher scores indicate greater balance confidence.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
score on a scale | 3.5 (0.4) | 3.2 (0.7)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); Test type: Superiority; p = 0.005, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

22. Secondary Outcome: Activities-Specific Balance Confidence Scale (ABC), Participants With Bilateral Amputation
Description: as for outcome 21
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
score on a scale | 3.4 (0.3) | 3.0 (0.5)

23. Secondary Outcome: Trinity Amputation Prosthesis Experience Scales, Revised (TAPES-R), Participants With Unilateral Amputation
Description: The TAPES-R is a self-report instrument designed to evaluate respondent's activity restrictions and satisfaction with a prosthesis. The TAPES-R has three subscales (activity restrictions [TAPES-AR], functional satisfaction [TAPES-FUN], and aesthetic satisfaction [TAPES-AES], each scored from 0 to 2. Higher scores indicate more activity restrictions (TAPES-AR) or greater satisfaction (TAPES-FUN and TAPES-AES). Participants were administered an electronic version of the TAPES-R on an iPad tablet.
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mRSF (Unilateral) | ESF (Unilateral)
Number analyzed (Participants) | 27 | 27
score on a scale
  TAPES-AR | 0.4 (0.3) | 0.6 (0.4)
  TAPES-FUN | 1.8 (0.4) | 1.3 (0.5)
  TAPES-AES | 1.5 (0.5) | 1.5 (0.5)
Statistical Analysis 1: Comparison: mRSF (Unilateral) vs ESF (Unilateral); TAPES-AR results; Test type: Superiority; p = 0.002, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05
Statistical Analysis 2: Comparison: mRSF (Unilateral) vs ESF (Unilateral); TAPES-FUN results; Test type: Superiority; p < 0.001, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05
Statistical Analysis 3: Comparison: mRSF (Unilateral) vs ESF (Unilateral); TAPES-AES results; Test type: Superiority; p = 0.85, t-test, 2 sided — Holm-Bonferroni adjustments for multiple comparisons were applied to yield an experiment-wise alpha level of .05

24. Secondary Outcome: Trinity Amputation Prosthesis Experience Scales, Revised (TAPES-R), Participants With Bilateral Amputation
Description: as for outcome 23
Time Frame: Participants were tested after using each foot in their prosthesis for 1 month.
Population: Data are from participants with bilateral amputation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mRSF (Bilateral) | ESF (Bilateral)
Number analyzed (Participants) | 5 | 5
score on a scale
  TAPES-AR | 0.7 (0.2) | 0.9 (0.2)
  TAPES-FUN | 1.8 (0.4) | 1.1 (0.2)
  TAPES-AES | 1.8 (0.3) | 0.9 (0.5)

ADVERSE EVENTS:
Time Frame: One month for each intervention
Description: All participants who received at least one intervention (prosthetic foot)
Groups:
- mRSF (Unilateral and Bilateral): Participants with unilateral and bilateral amputation tested while wearing the mRSF.
- ESF (Unilateral and Bilateral): Participants with unilateral and bilateral amputation tested while wearing the ESF.
Arm/Group | mRSF (Unilateral and Bilateral) | ESF (Unilateral and Bilateral)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2015-02-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT02440711/Prot_ICF_000.pdf